CLINICAL TRIAL: NCT03309826
Title: Effects of Positive Airway Pressure Treatment of Obstructive Sleep-disordered Breathing on Maternal and Fetal Outcomes in Hypertensive Disorders of Pregnancy: a Pilot Randomized Controlled Trial
Brief Title: Positive Airway Pressure Treatment of Obstructive Sleep-disordered Breathing in Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr John Kimoff (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); ResMed Canada Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Dr John Kimoff, Professor of Medicine, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-2856
Record Dates: First submitted 2017-09-25; First posted 2017-10-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hypertensive Disorder of Pregnancy; Sleep Apnea, Obstructive
Keywords: gestational hypertension; pre-eclampsia; eclampsia; obstructive sleep apnea-hypopnea; positive airway pressure; polysomnography; blood pressure; arterial stiffness
MeSH Terms: conditions — Toxemia; Sleep Apnea, Obstructive; Hypertension, Pregnancy-Induced; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analysis of all outcome measures will be conducted on a blinded basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAP Treatment Arm (Experimental): Automated positive airway pressure titration then treatment with fixed PAP.
  Interventions: Device: Positive Airway Pressure
- Nasal Dilator Strip (Active Comparator): Nightly use of nasal dilator strip
  Interventions: Device: Nasal Dilator Strip

INTERVENTIONS:
Device: Positive Airway Pressure — Auto-PAP titration followed by fixed PAP treatment
  Other Names: PAP
  Arms: PAP Treatment Arm
Device: Nasal Dilator Strip — Nightly use of nasal dilator strip
  Arms: Nasal Dilator Strip

SUMMARY:
The purpose of this study is to conduct a pilot randomized, controlled trial to evaluate the feasibility and obtain pilot outcome data for a subsequent definitive trial evaluating the effects of postitive airway pressure (PAP) treatment of obstructive sleep-disordered breathing (OSDB) on blood pressure control and maternal and fetal outcomes in hypertensive disorders of pregnancy. The primary aim of the pilot study is to assess feasibility measured as the rates of subject recruitment, adequate (>4h/night) PAP adherence (primary outcome measure) and protocol completion. Secondary aims will be to obtain preliminary data on the effects of PAP on maternal blood pressure, complications of hypertension, arterial stiffness and vascular biomarkers, course of labor and delivery and fetal outcomes including growth restriction, prematurity, and neonatal distress.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 y with a singleton pregnancy, ≥ 12 weeks' gestation
* diagnosis of hypertensive disorder of pregnancy, including pre-existing hypertension, gestational hypertension and pre-eclampsia, as defined by Canadian Hypertensive Disorders of Pregnancy Working Group Criteria (Magee et al; Best Practice and Research Clinical obstetrics & Gynaecology. 2015;29(5):643-657)
* presence of obstructive sleep-disordered breathing (OSDB) on a single night in-home complete (Level 2) polysomnogram defined by an apnea-hypopnea index (AHI) ≥ 5 events/h and/or the presence of inspiratory flow limitation on ≥ 30% of breaths.

Exclusion Criteria:

* severe pre-eclampsia/eclampsia requiring urgent delivery
* chronic kidney disease or other secondary cause of hypertension
* known cardiac disease, transient ischemic attack/stroke
* malignancy or other chronic medical or psychiatric condition
* smoking, alcohol use, illicit drugs
* current/recent treatment for sleep-disordered breathing
* severe sleep-disordered breathing defined as an apnea-hypopnea index (AHI) ≥ 30/h with either severe sleepiness (Epworth sleepiness score ≥ 15) or hypoxemia (4% Oxygen Desaturation Index ≥30/h or arterial oxygen saturation (SpO2) <80% for >10% of Total Sleep Time)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender defined by pregnancy
Enrollment: 48 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PAP Adherence | Through study completion, 8 weeks post-partum
  The proportion of subjects demonstrating >4h/night CPAP use by objective; microprocessor monitoring

SECONDARY OUTCOMES:
Subject recruitment rates | Through study completion, 8 weeks post-partum
  Percent recruitment of eligible subjects
Subject retention rates | Through study completion, 8 weeks post-partum
  Number of subjects completing the study protocol
Maternal 24 hour blood pressure | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  24 hour ambulatory blood pressure
Maternal blood pressure | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  Standardized blood pressure measurements using "BPTru" device
Arterial stiffness measured as carotid-femoral pulse wave velocity | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  Non-invasive measurement of arterial stiffness using applanation tonometry
Epworth Sleepiness Score | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  Standard subjective sleepiness score
Pittsburgh Sleep Quality Index | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  Subjective sleep quality index
Restless leg syndrome questionnaire | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  International Restless Legs Study Group questionnaire
Functional Outcomes of Sleep Questionnaire | Baseline, approximately one week prior to delivery and 8 weeks post-partum
  Sleep-related quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John Kimoff, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smocot J, Huynh N, Panyarath P, Kimoff RJ, Meltzer S, Drouin-Gagne L, Newbold R, Hebert C, Benedetti A, Arcache JP, Morency AM, Garfield N, Rey E, Pamidi S. Patterns of adherence to continuous positive airway pressure and mandibular advancement splints in pregnant individuals with sleep-disordered breathing. Sleep Breath. 2025 Apr 4;29(2):148. doi: 10.1007/s11325-025-03284-5. PMID 40183988
- [Derived] Panyarath P, Goldscher N, Pamidi S, Daskalopoulou SS, Gagnon R, Dayan N, Raiche K, Olha A, Geater SL, Benedetti A, Kimoff RJ. Positive Airway Pressure Treatment of Obstructive Sleep Apnea-Hypopnea in Hypertensive Disorders of Pregnancy: A Pilot Randomized Proof-of-Concept Clinical Trial. Ann Am Thorac Soc. 2024 May;21(5):803-813. doi: 10.1513/AnnalsATS.202310-863OC. PMID 38252423